CLINICAL TRIAL: NCT07019870
Title: Screening for Early Diagnosis of Nose Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); Genome Institute of Singapore (Other); Pathnova Laboratories, Singapore (Unknown); National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2022/00507
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Community screening; EBV IgA serology; Plasma EBV DNA
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Masking Description: Laboratories performing the EBV EA IgA serology and plasma EBV DNA are blinded to the clinical outcome of the participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Risk Individuals (Other): High risk individuals are determined by:
  a positive EBV EA IgA serology test, and/or two consecutive positive plasma EBV DNA tests
  High risk individuals will undergo evaluation in the outpatient Otolaryngology clinic. The evaluation includes a head and neck examination, nasoendoscopy and nasopharyngeal biopsy. Clinical data will be collected at yearly intervals, for at least 3 years, with annual clinical examination and blood tests.
  Interventions: Diagnostic Test: EBV biomarker testing
- Low Risk Individuals (Other): Low risk individuals are determined by: a negative EBV EA IgA serology, and negative plasma EBV DNA test (i.e. a negative plasma EBV DNA test, or an initially positive plasma EBV DNA test followed by a negative plasma EBV DNA test on repeat blood taking).
  Low risk individuals will be contacted via phone call every year for at least 3 years to confirm their disease status. Records will also be reviewed at the National Registry of Disease Office, to confirm that the participant has not been diagnosed with NPC.
  Interventions: Diagnostic Test: EBV biomarker testing

INTERVENTIONS:
Diagnostic Test: EBV biomarker testing — 15 ml of blood will be collected for EBV EA IgA serology and plasma EBV DNA testing by a trained nursing/phlebotomy staff. If the initial plasma EBV DNA test is positive, a second blood draw will be performed for repeat plasma EBV DNA testing.
  Additionally, 2-3 ml of saliva will be collected for EBV strain identification, however, this information is not used for risk stratification in this study.
  Demographic characteristics, clinical history and symptoms will be collected through a questionnaire.

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of screening in identifying nasopharyngeal cancer (NPC), and evaluate the performance of Epstein-Barr virus (EBV) biomarkers in a community screening setting in Singapore.

Participants will assessed for their risk of NPC using EBV Early Antigen (EA) IgA serology and cell-free plasma EBV DNA. If the initial plasma EBV DNA test is positive, a repeat blood sample will be taken and tested. Saliva will also be collected for evaluation of EBV risk strains, but not used for risk evaluation.

1. High risk individuals are determined by:

   * a positive EBV EA IgA serology test, and/or
   * two consecutive positive plasma EBV DNA tests

   High risk individuals will undergo evaluation in the outpatient Otolaryngology clinic. The evaluation includes a head and neck examination, nasoendoscopy and nasopharyngeal biopsy. Clinical data will be collected at yearly intervals, for at least 3 years, with annual clinical examination and blood tests.
2. Low risk individuals are determined by:

   * a negative EBV EA IgA serology, and
   * a negative plasma EBV DNA test, or an initially positive plasma EBV DNA test followed by a negative plasma EBV DNA test on repeat blood taking.

Low risk individuals will be contacted via phone call every year for at least 3 years to confirm their disease status. Records will also be reviewed at the National Registry of Disease Office, Health Promotion Board, to confirm that the participant has not been diagnosed with nasopharyngeal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Chinese, Malay, and mixed ethnicities
* individuals not diagnosed with NPC
* individuals with family history of NPC

Exclusion Criteria:

* younger than 35, older than 60
* individuals already diagnosed with NPC
* pregnant women

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male (n = 15,000) and female (n = 5000)
Enrollment: 20000 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Stage distribution of NPC | From enrollment of the participant to follow-up at three years
  Stage distribution of NPC diagnosed in study participants, compared to stage distribution of NPC in unscreened individuals routinely diagnosed in the clinic.
Accuracy of EBV IgA serology in identifying NPC cases | From enrollment of the participant to follow-up at three years
  Accuracy of EBV IgA serology including sensitivity, specificity, positive predictive value and negative predictive value
Accuracy of plasma EBV DNA in identifying NPC cases | From enrollment of the participant to follow-up at three years
  Accuracy of plasma EBV DNA including sensitivity, specificity, positive predictive value and negative predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Kwok Seng Loh, MBBS, FRCS, Principal Investigator — National University Health System, Singapore; Joshua K Tay, MBBS, PhD, Principal Investigator — National University Health System, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - National University Polyclinics, Singapore

IPD SHARING:
Plan to Share IPD: Undecided